CLINICAL TRIAL: NCT07210346
Title: The Effects of Listening to Fairy Tales, Listening to Fairy Tales in Their Mothers' Voices, and Watching Cartoons on Pain, Comfort Levels, and Physiological Parameters During Tracheostomy Care in a Palliative Care Clinic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Fatma Güdücü Tüfekci, Prof. Dr., Ataturk University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pediatric Nursing
Record Dates: First submitted 2025-09-10; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Tracheostomy; Care
Keywords: Palliative care; Children; Listening to stories; Watching Cartoons; Pain; Comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine tracheostomy care will be applied to the control group. No action will be taken.
- Experimental Group (Experimental): During the tracheostomy care process, the experimental group will listen to fairy tales and watch cartoons.
  Interventions: Other: fairy tales; Other: mother's voice; Other: Cartoons

INTERVENTIONS:
Other: fairy tales — The children's stories will be selected by child psychologists. The stories will be read by a story therapist and recorded on a voice recorder. The story playback will begin five minutes before the request begins and continue throughout the request process. The stories will be played for five days. Afterward, there will be a one-week detoxification period before moving on to the next intervention.
  Arms: Experimental Group
Other: mother's voice — Children's stories will be selected by child psychologists. The stories will be read by the children's mothers and recorded on a voice recorder. Story repetition will begin five minutes before the request begins and continue throughout the request period. The stories will be listened to for five days. Following this, there will be a one-week detoxification period before moving on to the next intervention.
  Arms: Experimental Group
Other: Cartoons — The cartoons children will watch will be selected by child psychologists. Children will be shown cartoons on tablets. Watching will begin five minutes before the request period and continue throughout the request period. Children will be shown cartoons for five days.
  Arms: Experimental Group

SUMMARY:
This study aimed to determine the effects of listening to fairy tales, listening to fairy tales from the mother's voice, and watching cartoons on pain, comfort, and physiological parameters during tracheostomy care of children receiving palliative care.

DETAILED DESCRIPTION:
Seventeen volunteer children between the ages of 1 and 7 receiving palliative care will be randomly assigned to three groups: a storytelling group, a mother's voice storytelling group, and a cartoon group. Each intervention will be administered once a day for one week. There will be a one-week washout period between interventions, during which time the children will receive routine nursing care. No intervention other than the storytelling or cartoon intervention will be administered to all three groups. Children will be assessed before, during, and after the procedure. PAIN RELATED TO THE TRACEOSTOMY PROCEDURE will be assessed using the FLACC Pain Scale, and comfort will be assessed using the Child Comfort Scale. Additionally, the children's heart rate, respiration, blood pressure, tidal volume, and temperature will be measured using a bedside monitor.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 1-7 year old age group,
* Being inpatient in a pediatric palliative care unit,
* Having no visual or hearing abnormalities,
* Having a tracheostomy.

Exclusion Criteria:

* The family's desire to withdraw from the study,
* The child's health condition deteriorates.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
FLACC Pain Scale | baseline and up to 1 weeks
  FLACC has reliability and validity to determine observational pain of children aged between 3 and 18 years during the medical procedures. This scale is preferred due to its implicity of application among children. It has five categories of behavior to rate pain, namely, facial expression, leg movement, activity, cry, and consolability. The scores of each category are between 0 and 2. The total scores can range from 0 to 10, defined as mild (1-3), moderate (4-6), and severe (7-10). The higher the score, the greater the pain.
Comfort Scale | baseline and up to 1 weeks
  It is a sedation and comfort scoring system that includes two physiological and six emotional stress criteria. While it assesses sedation patterns in ventilated children, the parameters assessed can also be considered indicators of pain. The patient child is assessed on six behavioral parameters (alertness, calmness-agitation, respiratory response, physical movement, muscle tone, and facial tension) and two physical parameters (blood pressure and heart rate) within two minutes. Each criterion is scored on a Likert-type scale from one to five. The assessment result is: 27-40 indicates light sedation, 17-26 indicates moderate sedation, and 8-16 indicates deep sedation. The comfort scale assesses the child's level of sedation and also influences pain and comfort levels.

SECONDARY OUTCOMES:
Patient Identification Form | Baseline Characteristics
  In this form, there are questions about the child's age, gender, diagnosis of the disease, length of stay, and how long ago she received the current diagnosis.
Physiological Parameter Record Form | Baseline and up to 1 week
  In this form, there are records of all physiological parameters including pulse and respiratory rate, body temperature, blood pressure, SpO2, tidal volume, and peak heart rate. If the value of each parameter is higher than the normal values, it indicates the presence of abnormal condition. Pulse normal value range: 80-130/ Minute Blood pressure normal value range:92-44 mmHg Respiratory rate normal value range: 16-22/ Minute Body temperature normal value range: 36,4-38 degree SpO2 normal value range: %96-98 Tidal volume normal value range: 6-10 ml/kg

CONTACTS AND LOCATIONS:
Overall Officials: Fatma GÜDÜCÜ TÜFEKCİ, 1, Study Chair — Ataturk University
Locations (1):
- Erzurum City Hospital, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarialioglu A, Kurudirek F, Oluc T. The effect of storybook reading on children's preoperative fear and anxiety levels: A randomized controlled study. Child Care Health Dev. 2023 Sep;49(5):906-913. doi: 10.1111/cch.13100. Epub 2023 Feb 8. PMID 36735635
- See also: Randomized Controlled Trial — http://pubmed.ncbi.nlm.nih.gov/36735635/